CLINICAL TRIAL: NCT01437735
Title: A Randomized, Placebo-controlled, Dose-ranging, Multi-centre Trial of QAW039 (1-450 mg p.o.), to Investigate the Effect on FEV1 and ACQ in Patients With Moderate-to-severe, Persistent, Allergic Asthma, Inadequately Controlled With ICS Therapy.
Brief Title: Dose Finding Study for QAW039 in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAW039A2206; 2011-001062-18 (EudraCT Number)
Record Dates: First submitted 2011-09-14; First posted 2011-09-21 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: Asthma; QAW039
MeSH Terms: conditions — Asthma | interventions — fevipiprant; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (15):
- QAW039 po dose 1 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 2 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 3 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 4 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 5 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 6 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 7 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 8 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 9 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 10 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 11 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 12 (Experimental)
  Interventions: Drug: QAW039
- QAW039 po dose 13 (Experimental)
  Interventions: Drug: QAW039
- Montelukast po 10 mg (Active Comparator): Comparator leukotriene receptor antagonist (LRTA)
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039 — QAW039 po
  Arms: QAW039 po dose 1; QAW039 po dose 10; QAW039 po dose 11; QAW039 po dose 12; QAW039 po dose 13; QAW039 po dose 2; QAW039 po dose 3; QAW039 po dose 4; QAW039 po dose 5; QAW039 po dose 6; QAW039 po dose 7; QAW039 po dose 8; QAW039 po dose 9
Drug: Montelukast — Montelukast 10 mg po
  Arms: Montelukast po 10 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to demonstrate a clinically significant improvement in Forced Expiratory Volume in one second (FEV1) in moderate to severe allergic asthmatics inadequately controlled by Inhaled Corticosteroid (ICS) therapy. Patients will be treated with QAW039, an active comparator, or placebo. This will be a randomized, placebo-controlled, dose-ranging, multi-centre trial.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma, as per the Global Initiative for Asthma (GINA) (2009) guidelines, and currently prescribed Inhaled Corticosteroids (ICS) therapy.
* Patients with a pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1) value of 40% to 80% of individual predicted value.
* Patients should be allergic or atopic, as diagnosed historically or prior to entry into the study.
* Patients who are demonstrated to have reversible airway obstruction or airways hyper-reactivity or have shown either of such responses in previous test(s) within the last year.
* An Asthma Control Questionnaire (ACQ) score ≥ 1.5 at randomization.

Exclusion Criteria:

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/mL).
* Patients with serious co-morbidities including uncontrolled diabetes (HbA1c≥8%), heart failure, cancer, neurodegenerative diseases, rheumatoid arthritis and other autoimmune diseases, other lung diseases including chronic bronchitis, chronic obstructive pulmonary diseases or emphysema or other conditions characterized by eosinophilia and pulmonary symptoms (i.e. Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis, eosinophilic pneumonia, etc.).
* Acute illness other than asthma at the start of the study
* History of life-threatening asthma, including a history of significant hypercarbia (pCO2>45mmHg), prior intubation, respiratory arrest, or seizures as a result of asthma.
* Patients who have had a respiratory tract infection within 4 weeks of the screening visit. Patients who develop a respiratory tract infection between screening and the randomization visit must be screen failed, and may be permitted to re-enroll at a later date.
* Current smokers or ex-smokers who stopped smoking within 6 months prior to screening or have a smoking history of ≥ 10 pack years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1043 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in trough Forced Expiratory Volume in 1 second (FEV1) from baseline to week 12 | Baseline and week 12
  Forced Expiratory Volume in 1 second (FEV1) (measured in litters), and the trough measurement is taken 24 hours after morning dose on the previous day.

SECONDARY OUTCOMES:
Change in Asthma Control Questionnaire (ACQ) score from baseline to week 12 | Baseline and week 12
  The Asthma Control Questionnaire (ACQ) is a validated questionnaire consisting of 7 items: 5 on symptom assessment, 1 on rescue bronchodilator use and 1 assessing the patients Forced Expiratory Volume in 1 second (FEV1) result against the predicted result for a person of similar age and stature. Each item is graded on a scale of 0-6, and a mean score of 1.5 or greater is considered to demonstrate inadequate asthma control in this trial. The minimal important difference that is considered clinically important is a change of 0.5 in the mean score.
Change in Forced Expiratory Volume in 1 second (FEV1) from baseline to weeks 2, 4 and 8. | Baseline, week 2, week 4 and week 8
  Forced Expiratory Volume in 1 second (FEV1) (measured in litters), and the measurement is taken 24 hours after the morning dose on the previous day.
Change in the Asthma Control Questionnaire (ACQ) score from baseline to weeks 2, 4 and 8. | Baseline, week 2, week 4 and week 8
  The Asthma Control Questionnaire (ACQ) is a validated questionnaire consisting of 7 items: 5 on symptom assessment, 1 on rescue bronchodilator use and 1 assessing the patients Forced Expiratory Volume in 1 second (FEV1) result against the predicted result for a person of similar age and stature. Each item is graded on a scale of 0-6, and a mean score of 1.5 or greater is considered to demonstrate inadequate asthma control in this trial. The minimal important difference that is considered clinically important is a change of 0.5 in the mean score.
Change in the dose response relationship among QAW039 doses with respect to Forced Expiratory Volume in 1 second (FEV1) after 12 weeks treatment. | Baseline and week 12
  Forced Expiratory Volume in 1 second (FEV1) (measured in litters), and the measurement is taken 24 hours after the morning dose on the previous day.
Comparison of vital signs, ECG, laboratory tests and adverse events across QAW039 doses and placebo. | Baseline and week 12
  Comparisons of vital signs (i.e. systolic and diastolic blood pressure, pulse rate), ECG (e.g. quantitative assessments - heart rate, QTcF, PRS, PR intervals), laboratory tests (haematology, clinical chemistry and urinalysis) and adverse events across QAW039 doses and placebo.
Comparison of efficacy of QAW039 with that of active comparator as an add-on therapy to Inhaled Corticosteroids (ICS) | Baseline and week 12
  Forced Expiratory Volume in 1 second (FEV1) measurement taken 24 hours after the morning dose on the previous day. The Asthma Control Questionnaire (ACQ)consisting of 7 items: 5 on system assessment, 1 on rescue bronchodilator use and 1 assessing the patients for FEV1 result against the predicted result for a person of similar age and stature. Each item is graded on a scale of 0-6, and a mean score of 1.5 or greater is considered to demonstrate inadequate asthma control in this trial. The minimal important difference that is considered clinically important is a change of 0.5 in the mean score.
Assess the effect of QAW039 on asthma symptoms as measured by asthma control diary. | Baseline and week 12
  The asthma control diary mimics the Asthma Control Questionnaire (ACQ), but is recorded daily by the patient, rather than at each visit. As for the ACQ, the ACD consists of 7 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (181):
- United States (36):
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Encinitas, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, San Mateo, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Centennial, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, River Forest, Illinois
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Wheaton, Maryland
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Warrensburg, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Papillion, Nebraska
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Lake Oswego, Oregon
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Lincoln, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Waco, Texas
  - Novartis Investigative Site, South Burlington, Vermont
- Argentina (9):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, San Juan Bautista, Buenos Aires
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Santa Fe
- Austria (5):
  - Novartis Investigative Site, Feldbach
  - Novartis Investigative Site, Grieskirchen
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Thalheim bei Wels
  - Novartis Investigative Site, Vienna
- Bulgaria (4):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (3):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Québec, Quebec
- Colombia (5):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Armenia
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Medellín
- France (8):
  - Novartis Investigative Site, Ferolles-Attily, France
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Tarbes
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Heraklion - Crete, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Guatemala (2):
  - Novartis Investigative Site, Antigua Guatemala
  - Novartis Investigative Site, Guatemala City
- Hungary (8):
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Deszk
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Mosonmagyaróvár
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Százhalombatta
  - Novartis Investigative Site, Törökbálint
- India (12):
  - Novartis Investigative Site, Panjim, Goa
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Nagpur - Maharashtra, India
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Indore, Madhya Pradesh
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
- Italy (3):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Parma, PR
- Japan (40):
  - Novartis Investigative Site, Nishio, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Mizunami, Gifu
  - Novartis Investigative Site, Hatsukaichi, Hiroshima
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Higashiibaraki-gun, Ibaraki
  - Novartis Investigative Site, Hitachi, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Tsukubo-gun, Okayama-ken
  - Novartis Investigative Site, Habikino, Osaka
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Tachikawa, Tokyo
  - Novartis Investigative Site, Taitō City, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kochi
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Osaka
- Mexico (5):
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- Netherlands (2):
  - Novartis Investigative Site, Almelo
  - Novartis Investigative Site, Harderwijk
- Peru (6):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, Miraflores, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, Santiago de Surco, Lima region
- Poland (2):
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
- Romania (7):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Iași, Jud. Iasi
  - Novartis Investigative Site, Arad
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Deva
- Russia (6):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- South Africa (7):
  - Novartis Investigative Site, Benoni
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, eManzimtoti
  - Novartis Investigative Site, Gatesville
  - Novartis Investigative Site, Port Elizabeth
  - Novartis Investigative Site, Pretoria
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Yenisehir/Izmir
- United Kingdom (3):
  - Novartis Investigative Site, Newcastle upon Tyne, Newcastle
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Glasgow - Scotland

REFERENCES:
- [Derived] Bateman ED, Guerreros AG, Brockhaus F, Holzhauer B, Pethe A, Kay RA, Townley RG. Fevipiprant, an oral prostaglandin DP2 receptor (CRTh2) antagonist, in allergic asthma uncontrolled on low-dose inhaled corticosteroids. Eur Respir J. 2017 Aug 24;50(2):1700670. doi: 10.1183/13993003.00670-2017. Print 2017 Aug. PMID 28838980
- See also: Results for CQAW039A2206 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13023